CLINICAL TRIAL: NCT05978531
Title: A Prospective, Observational Study of Bafiertam Evaluating Persistence on Treatment, Safety, Tolerability, and Effectiveness in Routine Clinical Practice.
Brief Title: Observational Study of Persistence on Bafiertam Treatment in Routine Clinical Practice
Acronym: SIMPLE
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Banner Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BLS-11-404
Record Dates: First submitted 2023-07-25; First posted 2023-08-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — monomethyl fumarate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Monomethyl Fumarate — 95 mg oral capsule, 190 mg (2 x 95 mg) twice daily
  Other Names: Bafiertam; BLS-11

SUMMARY:
This is an open-label, multicenter, observational study of the adherence of patients with relapsing-remitting multiple sclerosis (RRMS) prescribed Bafiertam (monomethyl fumarate) as their treatment.

DETAILED DESCRIPTION:
Monomethyl fumarate (MMF) is the active metabolite of the fumarate class of drugs used for the treatment of RRMS. Bafiertam is a formulation of MMF and does not require enzymatic conversion after oral administration. Adult participants with a diagnosis of RRMS who have been receiving continuous treatment with Bafiertam monotherapy per the approved product label for no more than 3 months (90 days) are eligible to enroll in the study. Their satisfaction with Bafiertam treatment will be assessed using a 9-Item Treatment Satisfaction Questionnaire for Medication (TSQM-9). To be included in the study, patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged 18 years and older.
2. Participants diagnosed with Relapsing forms of multiple sclerosis R(RMS) and satisfy the approved therapeutic indication for Bafiertam per the approved product labeling.
3. Participants may enroll if they are within 90 days of initiating therapy with Bafiertam.
4. Female participants of childbearing potential must practice effective contraception from Day -1 and be willing and able to continue contraception for the duration of the study.
5. Willing and able to sign the informed consent form (ICF) approved by the Institutional Review Board (IRB).
6. Willing and able to complete all the study procedures and communicate meaningfully with study personnel.

Exclusion Criteria:

1. Known hypersensitivity to fumarates including dimethyl fumarate, Tecfidera, and/or diroximel fumarate (Vumerity) or Bafiertam.
2. Participated in another clinical trial within 30 days, suffered or still recovering from a medically significant event of surgery within 30 days, or previously participated in a clinical study with a similar investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from existing patients known to the individual investigators.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Percentage of participants on treatment with Bafiertam at 1 Year. | 12 months
  Percentage of participants on treatment with Bafiertam at 1 Year.

SECONDARY OUTCOMES:
Percentage of Participants on Treatment with Bafiertam at 6 months | 6 months
  Percentage of Participants on Treatment with Bafiertam at 6 months
Treatment Satisfaction Questionnaire for Medication (TSQM-9) | 12 months
  Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9) Total Score (range 0 - 100) at Month 6 and 12 months.TSQM Version 9 is comprised of 9 questions that provide scores on four scales: effectiveness (3 items), convenience (3 items), and global satisfaction (3 items). The scale scores are transformed and range from 0 to 100. Higher scores indicate greater satisfaction.
Number of Participants with Adverse Events (AEs) Leading to Treatment Discontinuation. | 12 months
  Number of Participants with AEs Leading to Treatment Discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lategan, PhD, Study Director — Banner Life Sciences
Locations (10):
- United States (9):
  - Gilbert Neurology, Gilbert, Arizona
  - Center for Neurology and Spine, Phoenix, Arizona
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Clinical Endpoints, Scottsdale, Arizona
  - Regina Berkovich MD PhD Inc., West Hollywood, California
  - Comprehensive Neurology Clinics of Bethesda Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Maryland Center for Neurology and Sleep, Glen Burnie, Maryland
  - Holy Name Medical Center, Teaneck, New Jersey
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Caribbean Center for Clinical Research/San Juan MS Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No